CLINICAL TRIAL: NCT04442568
Title: Enhanced Recovery After Surgery Protocol in Laparoscopic Sleeve Gastrectomy
Brief Title: Impact of ERAS in LSG
Acronym: ERAS-LSG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Abdullah Sisik, Assoc. Prof., Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ERAS-LSG
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Laparoscopic Sleeve Gastrectomy; Enhanced Recovery After Surgery; Pain, Postoperative; Nausea, Postoperative; Vomiting, Postoperative
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: Patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS (Active Comparator): all patients in this group will be performed LSG under a specified anesthesia protocol. This protocol includes non-opioid analgesia and sedation. Also short-acting anesthetic drugs will be used in this arm. The patients in this arm will be mobilized in the second hour postoperatively, also will be started oral intake between second and fourth hours.
  Interventions: Other: ERAS
- no ERAS (No Intervention): all patients in this group will be performed LSG under a conventional anesthesia protocol which is depended on the anesthesiologist . This protocol includes opioid analgesia and sedation. Also short and long acting anesthetic drugs will be used in this arm. The patients in this arm will be mobilized in the fourth hour postoperatively, also will be started oral intake in the next day morning after surgery.

INTERVENTIONS:
Other: ERAS — early mobilisation, early oral intake, early discharge
  Arms: ERAS

SUMMARY:
Patients with BMI >35 and chronic diseases or BMI >40 will be scheduled to receive Laparoscopic Sleeve Gastrectomy (LSG). Two groups are planned according to receive Enhance recovery after surgery (ERAS) protocol or not. All participants will receive standard LSG. Participants of ERAS will receive anesthesia and post-surgical nutrition protocol which are determined for ERAS. All patients will be checked for status of pain with VAS score, nausea and vomiting with PONV score at postoperative 2nd hour, 12th hour. In ERAS group liquid oral intake will be started between postoperative 2nd and 4th hours. In no ERAS group liquid oral intake will be started in the morning of postoperative first day. The patients who provides discharge criterias will be discahrged. these criterias are; To provide adequate pain relief with paracetamol and nonsteroidal painkillers, No wound problem, No complications after surgery, Pulse rate <90 beats / min, temperature ≤ 37 · 5 ° C, respiratory rate, <20 breaths / minute, To be able to mobilize easily, To be able to drink 1 liter of water after surgery.

Emergency admissions of the participants within a month after surgery will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* must be performed laparoscopic sleeve gastrectomy
* body mass index > 35 with a comorbidıty or ,body mass index > 40

Exclusion Criteria:

* surgery with peroperative complication
* revision surgery applications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
length of hospital stay | till discharge, an average of 36 hours
  the time (in hours) from the start of surgery to the discharge of patients in both groups
number of emergency re-admission after surgery | during postoperative first 30 days
  number of emergency re-admission after surgery due to complications or patients discomfort
Score of Visual analog scale | postoperative 24 hours
  VAS scores that evaluate postoperative pain in both groups will be compared (minimum score 0, maxımum score 10 and higher scores mean a worse outcome)

REFERENCES:
- [Derived] Demirpolat MT, Sisik A, Yildirak MK, Basak F. Enhanced Recovery After Surgery Promotes Recovery in Sleeve Gastrectomy: A Randomized Controlled Trial. J Laparoendosc Adv Surg Tech A. 2023 May;33(5):452-458. doi: 10.1089/lap.2022.0494. Epub 2022 Dec 26. PMID 36576984